**Clinical Study Protocol** 



A prospective, randomized study comparing surgical and economic parameters of Total Knee Replacement performed using two different surgical techniques:

Medacta MyKnee® surgical technique using Efficiency single-use instruments versus Stryker Navigation surgical technique performed with conventional metal instruments.

# **Study Protocol**

Protocol #:

MyKnee-20170829

Sponsor:

Medacta USA, Inc,

Sponsor Contact:

Mukesh Ahuja, MBBS, MS, CCTI

Director of Clinical Research

1556 West Carroll Ave.

Chicago, IL 60607 Phone: 312-771-9615

Email: mahuja@medacta.us.com

## 1 INTRODUCTION

#### 1.1 STUDY RATIONALE

Total knee arthroplasties are a common procedure in the United States (US), designed to relieve pain and improve the quality of life in patients with advanced knee osteoarthritis. Age and obesity are major risk factors for osteoarthritis and as the US population continues to age and body mass index (BMI) levels increase, the incidence of total knee arthroplasties will increase as well. In 2013, total knee arthroplasties were occurring at a rate of greater than 500,000 procedures per Year and are expected to increase to 3.48 million by 2030.<sup>2</sup> Costs for total knee arthroplasties currently exceed \$11 billion in the US alone.<sup>1</sup>

With the numbers of total knee arthroplasties continuing to increase, efforts are being made to improve outcomes and to cut procedural costs. Accuracy of TKA placement is a key feature in providing for long term success, and is critical for limb alignment and knee biomechanics. Conventional TKA instrumentation has been the gold standard, yet other options are now available. To improve accuracy, TKA navigation systems have been developed and are evolving. many such systems require the use of sophisticated image tracking devices and bony reference pins, allowing for intraoperative data acquisition, analysis, and feedback to the surgeon regarding instrument placement. Studies have shown improved accuracy of navigation systems, but few have indicated long term outcome improvements in clinical performance and survivorship. For the same are also criticisms of navigation. Reference pins added to the femur and tibia can be sites of infection and/or stress fractures. Also, navigation is likely to add time to the procedure, raising concern for increased infection rates and costs. 11, 12, 13, 14

Another potential solution to increase accuracy and to decrease cost is patient-specific cutting blocks with single-use instruments. Patient-specific cutting blocks begin with preoperative imaging of the lower extremity alignment and knee, typically with CT or MRI, which is used to create 3-D digital models of the knee. The desired implant sizes and placement are optimized for individual knee anatomy and alignment, and this information is used to create patient-specific cutting blocks. These preclude the need for complex image acquisition devices and computers in the operating room. Such systems have been shown to decrease operative time, and no reference pins are needed in the femur or tibia. Furthermore, the utilization of single-use instruments can decrease the time spent preparing for and cleaning after the surgery, thereby decreasing patient turnover time.

Single-use instruments are common in ophthalmology, cardiothoracic surgery and urologic surgery, but have yet to experience much of a crossover into lower extremity surgery, including total joint arthroplasty. Mont et al. studied 400 procedures using single-use instruments for total knee arthroplasty, concluding that single-use instruments showed promising benefits and after further study, could play a role in increasing operating room efficiency.<sup>2</sup> Siegel et al. found that total operating room time during total knee arthroplasty was on average 30 minutes shorter for single-use instruments and saved between \$480 and \$600 per case.<sup>3</sup> The same study also suggested that single-use instrumentation may also decrease the risk of infection.

There is controversy regarding some manufacturers' claims of improved clinical outcomes, surgical efficiency and decreased costs with patient-specific cutting blocks. It is evident that not all patient-specific instruments from different manufacturers are equivalent, and each needs to be studied individually. This study is being conducted to compare the economic and clinical impact total knee replacement performed with patient-matched cutting blocks and single-use instrumentation versus navigation technique performed with conventional metal instrumentation.

## 1.2 STUDY TREATMENT

MyKnee® patient-specific cutting blocks allow the surgeon to realize his pre-operative 3D planning, based on CT images of the patient's knee. The blocks are created based on the individual patient's anatomy, his/her mechanical axis, and the surgeon's preferred reconstruction goals. The innovative concept combines the following features giving potential benefits to both the surgeon and the patient:

- Accurate bony cuts and therefore implant positioning
- No intramedullary canal violation
- Up to 60% reduction of surgical steps for bone resection and related time
- Up to 66% reduction of time and cost in washing, assembling and sterilization procedures
- Interactive 3D web planning

The GMK single-use (Efficiency) instruments are made of medical-grade composite technopolymers that give high fatigue and abrasion resistance in addition to form versatility. The single-use instruments are shipped from the manufacturer in pre-sterilized packaging, eliminating the need to use the hospital Central-Sterile processing equipment. The reproducible sterility may potentially reduce the infection risk.

## 1.3 STUDY OBJECTIVES

The objective of this research is to study the time-saving, economic and clinical impact of total knee replacement performed with patient-matched cutting blocks and single-use instrumentation versus navigation technique performed with conventional metal instrumentation.

#### Primary Objective:

- To compare the time-saving and economic parameters associated with the two procedures with respect to variables such as OR preparation time, intra-operative time (OR efficiency), OR clean-up time, cost of consumables, and sterilization costs.
- The cost-per-minute value based on hospital estimates will be used to calculate an overall cost-savings total.

#### Secondary Objectives:

To compare the following surgical and clinical outcomes between the two study groups

- To compare correction of alignment after total knee replacement via long standing AP hipknee-ankle x-rays.
- To compare the accuracy of tibial slope angle on a lateral knee x-ray
- To compare the number of trays sent to sterilization
- To compare the volume of estimated blood loss during the procedure
- To compare the drop in post-operative (day 1) hemoglobin and total volume of transfusions (allogeneic and/or autologous)
- To compare the occurrence of adverse events
- To compare the waste weight at the end of each surgery, considering separately those recyclable and those not recyclable.
- To compare the rate of intraoperative and post-operative complications
- To compare the rate of successful use of MyKnee® cutting blocks (i.e. the incidence of surgical cases where the surgeon did not need to abort the use of MyKnee intra-operatively and default to the use of standard cutting blocks or navigation technique.

## 2 STUDY DESIGN

The study is a prospective, randomized study comparing surgical and economic parameters of Total Knee Arthroplasty performed using two different patient specific surgical techniques: Medacta MyKnee® surgical technique using Efficiency single use instruments versus Stryker Navigation surgical technique performed with conventional metal instruments. The objective is to compare the impact of two different patient specific surgical techniques and instrumentation in reducing overall surgical costs and improving mechanical axis alignment in Total Knee Arthroplasty. The timing of routine surgical phases will be measured, including the pre-operative preparation time, intra-operative phase, OR clean-up time and sterilization phase in 134 adult patients undergoing total knee replacement. Long-standing (hip to ankle) AP and lateral x-rays will be utilized to assess the implant's mechanical axis alignment and tibial slope at 6 weeks post-op. Additionally, other parameters will be recorded including blood loss, post-op day 1 hemoglobin drop, adverse events, number of trays sent to sterilization, and total waste weight at the end of each procedure, considering separately those recyclable and those not recyclable. To ensure that the minimum of 134 patients is met, 150 patients will be randomized into two treatment cohorts in a 1:1 ratio.

Group A: Medacta MyKnee® Surgical Technique with Efficiency Single-Use Instruments
Patients randomized to Group A will undergo Total Knee Arthroplasty utilizing patient-matched cutting blocks (MyKnee®) and Efficiency single-use instrumentation.

**Group B: Stryker Navigation Surgical Technique with Conventional Metal Instruments**Patients randomized to Group B will undergo Total Knee Arthroplasty utilizing Stryker Navigation technology with conventional metal instrumentation.

Additional demographic information will be collected to describe the study population and to document whether the two treatment groups are clinically comparable. Data collected will include: age, gender, BMI, race/ethnicity, smoking history, and employment status, in addition to preoperative knee history/diagnosis and degree of pre-operative knee malalignment and Kellgren-Lawrence grade.

# 3 PATIENT RECRUITMENT AND SAMPLE SIZE

The study participants will be recruited from the patients receiving care with one of the study investigators or their practice partners. Participating clinicians and their staff will be notified of this protocol and will be asked to refer patients undergoing total knee arthroplasty.

150 patients will be enrolled and randomized to one of the two groups (n=75 for each group).

#### 3.1 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the investigator or qualified designee to ensure that the subject qualifies for the study prior to enrollment and randomization. Subjects must meet all inclusion criteria and none of the exclusion criteria to be eligible for the study.

## 3.1.1 Inclusion Criteria

In order to be eligible for participation in this study, the patient must meet all of the following inclusion criteria:

- 1) Age 18 to 75 years
- 2) BMI ≤35

- 3) Undergoing unilateral total knee arthroplasty due to osteoarthritis (primary or post-traumatic OA) with the Medacta GMK Sphere
- 4) Able and willing to give consent and to comply with study requirements, including follow up visit at 6 weeks

#### 3.1.2 Exclusion Criteria

The subject must be excluded from participating in the study if the subject meets any of the following exclusion criteria:

- 1) Is participating in another clinical study
- 2) Has inflammatory arthritis
- 3) Has knee avascular necrosis
- 4) Has severe deformity, defined as greater than 15 degrees varus or 10 degrees valgus relative to the mechanical axis.
- 5) Has retained hardware in the knee that requires removal and interferes with TKA procedure
- 6) Has prior high tibial osteotomy (HTO)

## 3.2 Study Procedures

Patients who are undergoing a unilateral total knee arthroplasty and meet all of the inclusion/exclusion criteria will be approached to participate in the study. If consent is obtained the study coordinator will be notified. The coordinator will randomize the patients in a 1:1 ratio to one of the two treatment cohorts (i.e., MyKnee® surgical technique with single use Efficiency Instrumentation or Stryker Navigation with conventional metal instrumentation). The study coordinator will notify the clinician of the treatment assignment. Subjects randomized to receive the MyKnee® surgical technique will have a CT scan and the investigator will perform appropriate pre-operative planning which enables the custom manufacturing of the MyKnee cutting blocks that will be delivered to the surgical facility. Subjects randomized to receive the Stryker Navigation surgical technique will not require CT scan. At the next visit the patient will undergo the total knee arthroplasty procedure utilizing the assigned instrumentation. Timing of various operative and sterilization phases will be recorded. Following the procedure, the patient will undergo X-rays at 6 weeks visit to examine the alignment of the implant.

## 3.2.1 Informed Consent

Individuals who agree to participate in this study will be asked to provide formal written informed consent. A signed copy of the informed consent form will be given to the patient, and the original will be maintained in the patient file.

Consent must be documented by the subject's dated signature or by the subject's legally acceptable representative's dated signature on a consent form along with the dated signature of the person conducting the consent discussion.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the subject must receive the IRB/EC's approval/favorable opinion in advance of use. The subject or his/her legally acceptable representative should be informed in a timely manner if new information becomes available that may be relevant to the subject's participation in the study. The communication of this information will be provided and documented via a revised consent form or addendum to the original consent form that captures the subject's dated signature or by the subject's legally acceptable representative's dated signature.

#### 3.2.2 Randomization

Patients will be randomized using a computer generated blocked randomization with equal allocation to the 2 different surgical techniques. The randomization will be performed separately for each site.

In case the investigator decides not to include the patient after randomization, this patient will be treated as withdrawn although a randomization has been performed. The reason for withdrawal must be documented in the patient file. The used randomization number cannot be used again. For the next patient, the following randomization number will be used.

#### 3.2.3 Protocol Deviations

Protocol deviations will be recorded and will capture the date of deviation, associated study visit, and type of deviation. Types of deviations are as follows:

- Consent procedures
- Inclusion/exclusion criteria
- Study procedures
- Serious adverse event / unanticipated adverse device effect (SAE/UADE) reporting
- Randomization procedures
- Visit schedule / window
- Other (site will be requested to specify)

## 3.3 EVALUATION PARAMETERS

### Time of Operative Phases

The time of the following pre-operative, operative and sterilization phases will be recorded (hh:mm:ss):

- 1. Surgery Room Preparation and Clean-up Phase
  - a. Instrument preparation for surgery from stock to Operative Room (OR)
  - b. Surgical table preparation
  - c. Instrument collection after surgery for sterilization
- 2. Intra-operative Phase
  - a. Patient OR time
  - b. Skin-to-skin time
  - c. Femoral and tibial resection times
  - d. Tourniquet time
- 3. Sterilization Phase
  - a. Instrument transportation to the sterilization unit
  - b. Instrument reception
  - c. Instrument cleaning before sterilization
  - d. Instrument decontamination before sterilization
  - e. Instrument sterilization
  - f. Instrument collection after sterilization
  - g. Instrument transportation to stock

#### Additional Operative Parameters

- 1. Estimated blood loss (cc)
- Drop in post-operative hemoglobin (measured at Day 1 or discharge if patient does not stay overnight)
- 3. Total volume of transfusions (allogeneic and/or autologous)
- 4. Number of trays sent to sterilization

5. Waste weight at the end of each surgery; recyclable and non-recyclable (grams)

## Radiographic Parameters

Each subject will undergo the following radiographic assessments pre-operatively and at 6 weeks post-operatively.

- Long standing (hip to ankle) AP x-ray to assess the mechanical axis alignment
- Standard lateral x-ray to assess tibial posterior slope

Accuracy will be determined by the difference between the final position on the post-operative x-rays and the surgeon's intended position (usually 0 degrees of mechanical axis on AP, and recreation of tibial slope on the lateral x-ray).

#### Adverse Events

All operative and post-operative adverse events, whether voluntarily reported by the patient or observed by the investigator, will be recorded in the patient's study records.

## 3.4 Study Visits

Each subject will attend 3 study visits. Each visit will have specified activities as described below.

## Visit 1: Baseline (-1 to -90 days prior to surgery)

The baseline visit will occur to screen subjects, confirm study eligibility, complete the informed consent process, and enroll and randomize the subject.

- Informed consent
- · Randomize patients meeting inclusion/exclusion criteria
- · Collect demographics data, pre-operative knee history/diagnosis and employment status
- Long standing (hip to ankle) AP and lateral x-rays to assess pre-operative mechanical axis alignment and posterior tibial slope. X-rays obtained within 6 months prior to surgery are acceptable for the baseline visit. The investigator may repeat x-rays if needed for clinical or imaging quality reasons.
- Complete CT scan for pre-operative planning and selection of cutting blocks (only for patients randomized to MyKnee Efficiency group)

## Visits 2: Operative (Day 0-Discharge)

The following activities will be performed at each surgery visit.

- · Surgery using instrumentation per randomization assignment
- Adverse event assessment
- Transfusion summary
- Bloodwork for hemoglobin assessment (measured at Day 1 or discharge if patient does not stay overnight)

# Visit 3: 6 Weeks (± 2 weeks)

The following activities will be performed at the post-operative/discharge visit.

- · Long standing (hip to ankle) AP x-ray to assess mechanical axis alignment
- Standard lateral x-ray to assess tibial slope
- · Adverse event assessment



| Activity | Baseline | Operative | 6 Weeks |
|---|---|---|---|
| Informed Consent | Х | | |
| Baseline Details | X | | |
| - Medical History | i | | |
| - Eligibility Criteria | X | 1 | |
| - Demographics | X | 1 | |
| CT Scan for Pre-Operative Planning | X | | |
| (MyKnee Group only) | _ ^ | | |
| Randomization | X | | |
| Operative Details | | X | |
| - Timing for Pre-Operative Phase | | X | |
| - Timing for Intra-Operative Phase | | X 1 | |
| - Timing for Sterilization Phase | | X | |
| - Other Operative Parameters | | X | |
| Adverse Events | | X <sup>1</sup> | X <sup>1</sup> |
| Long Standing and Lateral Knee X-Rays | X | | X |

<sup>&</sup>lt;sup>1</sup>If applicable.

# 3.5 Case Report Forms

Case Report Forms (CRFs) are to be completed for all subjects.

All data is collected on study source documents and entered into the Case Report Forms by the Study Coordinator or delegated designee. All data will be reviewed for consistency and correctness with the protocol by the Investigator (or designee) and the Clinical Research Associate (CRA). All discrepancies requiring verification via an examination of the source documents will be sent to the study site for resolution or resolved during monitoring visits. During monitoring visits, the CRA will review all data, evaluate for completeness and have the site enter missing information and/or resolve errors. All entries, corrections and alterations are to be made by the responsible Investigator or his/her designee.

## 3.6 Study Documents

The following documents will be required by each site prior to activation:

- Signed protocol signature page
- Signed and dated written approval from the IRB of the protocol, informed consent form, and any applicable recruiting materials
- · Signed investigator's agreement
- Financial disclosure form
- Signed and dated Delegation of Authority log
- · Curriculum Vitae and medical licenses of applicable study staff

## 4 STATISTICAL ANALYSIS PLAN

The Sponsor will evaluate for non-inferiority based on economic factors and the rate of adverse events between the two groups. The Sponsor may conduct additional post-hoc analyses of the study data after study completion. These analyses may be done for the purposes of publication or in conjunction with additional data that may be available to Sponsor from other sources.

#### 4.1 DATA ANALYSIS

The objectives of this study are outlined in Section 1.3. For purposes of this study, economic outcomes of interest include the peri-operative time, intra-operative time (OR efficiency), and sterilization times as quantitative values. These outcomes will be subsequently used in comparative cost analyses. The secondary objectives are to assess the accuracy of mechanical axis alignment

and posterior tibial slope after total knee replacement, additional operative parameters, and adverse events.

Descriptive statistics, specifically means will be used to summarize the peri-operative, intraoperative and sterilization time data.

The primary objective will be met by comparing mean values of each of the time-saving parameters. The null hypotheses of no differences in mean values between re-usable (Navigation with Conventional) and single-use (MyKnee with Efficiency) devices will be tested using separate t-tests for two independent groups for each endpoint. A p-value of less than 0.05 will be considered significant for each endpoint. Endpoints with statistically significant differences are expected to contribute to expected cost differences to be determined in subsequent analyses.

Descriptive analyses as well as similar two-sample comparisons will be used to evaluate secondary measures.

# 4.2 Sample Size Analysis

Sample size for this study was determined on the basis of device group differences observed in the Mont et al 2013 study for four (related) but important health care utilization endpoints. The table below summarizes the data in Table 2 of Mont et al, but also provides a summary of the comparisons between single-use and re-usable pooling over whether or not navigation was employed. These data were used to approximate the expected effect size (standardized mean difference) comparing between single-use vs re-useable instruments. The sample sizes required for a two sample t-test to obtain 80%, 85%, and 90% power as a function of the observed pooled effect sizes were determined. The effect sizes were derived from the reported mean differences and p-values. The maximum sample size per group required to achieve at least 80% statistical power to reject the null hypothesis of equal group mean was determined across the four outcomes summarized in MontTable 2. This sample size was 67 per group or total N=134. This value was increased by 12% to N=150 to account for uncertainty in the estimated effect sizes, to account and to allow for additional analyses of economic outcomes. Therefore, 150 patients will be randomly allocated to each of the experimental arms of the study.

## Sample Size for Main Effect of Navigation vs. MyKnee Efficiency

| Da | Data from Mont et al. (2013) Table 2 | | | | | | | Sample size calculations | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Outcome | | Trac | litional | Single Use | | p-<br>value | SD<br>estimate<br>d from<br>p-value | Conservati<br>ve SD<br>estimate | Diff b/w Trad+Y es & Single- Use+N o | N per<br>group<br>for<br>80%<br>powe<br>r | 85% | 90 % |
| | Na<br>v. | Pts | Mean | Pts . | Mean | | | | | | | |
| Instrume | No | 96 | 36.61 | 95 | 33.56 | 0.002 | 6.82 | 10.49 | 5.44 | 59 | 67 | 78 |
| nt set-up<br>time | Ye<br>s | 97 | 39.00 | 10 | 35.96 | 0.042 | 10.49 | | | | | |
| Instrume<br>nt<br>cleanup | No | 96 | 16.43 | 95 | 13.59 | 0.001 | 5.96 | 13.44 | 11.37 | 22 | 26 | 30 |
| | Ye<br>s | 97 | 24.96 | 10<br>0 | 20.09 | 0.011 | 13.44 | | | | 920 | |
| | No | 96 | 53.04 | 95 | 47.15 | 0.001 | 12.37 | 16.87 | 16.81 | 16 | 19 | 22 |

| Combine<br>d setup +<br>cleanup | Ye<br>s | 97 | 63.96 | 10<br>0 | 56.05 | 0.001 | 16.87 | | | | , | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Surgical<br>Episode | No | 96 | 100.5 | 95 | 97.11 | 0.100 | 14.58 | 18.98 | 31.40 | 6 | 7 | 8 |
| time | Ye | 97 | 128.5 | 10 | 119.6 | 0.001 | 18.98 | 1 | | | | |

### Sample size based on the variability of the resulting HKA

Anderl W et al study: Mean HKA-deviation from the targeted neutral mechanical axis (CVI:  $2.2^{\circ} \pm 1.7^{\circ}$ ; PSI:  $1.5^{\circ} \pm 1.4^{\circ}$ ; p < 0.001), rates of outliers (CVI:  $22.2^{\circ}$ ; PSI:  $9.6^{\circ}$ ; p = 0.016).

## Sample size based on rates of outliers

If we consider the rate of non-outliers to be (100%-9.6% approx. = 90%) in both Navigation and MyKnee groups, then for 80% power to establish non-inferiority of non-outliers for the MyKnee group at non-inferiority margin of 12.5%, we need a sample size of n=72 in each group.

## Sample size based on Mean HKA

If we consider the standard deviation of HKA-PSI to be 1.4 in both Navigation and MyKnee groups, then for 80% power to establish non-inferiority of HKA for the MyKnee group at non-inferiority margin of 0.6, we need a sample size of n=68 in each group.

## 5 BENEFIT/RISK PROFILE

## 5.1 Potential Benefits

. The study will provide the initial data to understand the health economic impact and effectiveness of MyKnee® TKA surgical technique with Efficiency single-use instrumentation as opposed to the Stryker Navigation TKA surgical technique with conventional metal instrumentation

#### 5.2 Possible Risks

It is not expected that the possible risks will increase with the instrumentation options. All risks are anticipated with total knee replacement surgery and surgery in general. The following risks and discomforts may occur and are considered anticipated in connection with total knee arthroplasty procedures at the time of the operation:

- Complication from Anesthesia
- Allergic Reaction

Deep Vein Thrombosis

Hemorrhage (Bleeding)

- Immunologic ResponseVascular Damage
- Nerve Damage
- Pulmonary EmbolismFat Emboli Syndrome
- The following risks and discomforts may occur with reusable or single-use instrumentation:
- Instrument Breakage
- Instrument Malfunction
- Retention of foreign body

## 6 ADVERSE EVENTS

Adverse event collection will begin from the time of first incision. All medical events and conditions that occur prior to this time point are to be captured as pre-existing conditions in the patient's medical history. Adverse event collection will conclude at the completion of the final follow-up visit.

Observed and reported adverse events shall be recorded in the patient's study records and on the Adverse Event Form within 48 hours of the site becoming aware of each event, and must include the following information at minimum:

- Event Description
- Date of Onset
- Date of Resolution
- Severity (mild, moderate, severe)
- Seriousness
- Relationship to surgery (definitely, probably, possibly, unlikely, not related)
- Relationship to instrumentation (definite, probable, possible, unlikely, not related)
- Event treatment (e.g., none, non-drug therapy, medications, surgery)
- Outcome

Significant new information and updates will continue to be captured in the patient's records as they become available. The investigator will follow each subject who experiences an AE until the event resolves or no further improvement is expected. If the AE has not resolved by the time of the subject's completion, the AE will be listed as ongoing at the time of subject discontinuation.

# 6.1 Assessment of Severity

The severity of the adverse event is classified as mild, moderate or severe.

- Mild: Awareness of signs or symptoms, but easily tolerated and are of minor irritant type causing no loss of time from normal activities. Symptoms do not require therapy or a medical evaluation; signs and symptoms are transient.
- Moderate: Events introduce a low level of inconvenience or concern to the participant and may interfere with daily activities, but are usually improved by simple therapeutic measures; moderate experiences may cause some interference with functioning.
- Severe: Events interrupt the participant's normal daily activities and generally require systemic drug therapy or other treatment; they are usually incapacitating.

## 6.2 Relationship to Surgery/Instrumentation

The investigator will evaluate the relationship of the adverse event to the research intervention according to the following definitions. The term "treatment-related," as it pertains to adverse events, means that the event was or may have been attributable to the treatment, or that the treatment was or may have been a factor in an event, including those occurring as a result of malfunction, poor manufacture, inadequate labeling, or improper design.

## Definitely

The adverse event is clearly related to the research intervention: the adverse event has a temporal relationship to the administration of the research intervention, follows a known pattern of response, or is otherwise logically related to the intervention, and no alternative cause is present.

## Probably

The adverse event is likely related to the research intervention: the adverse event has a temporal relationship to the administration of the research intervention, follows a known or suspected pattern of response, or is otherwise logically related to the intervention, but an alternative cause may be present.

Possibly

The adverse event may be related to the research intervention: the adverse event has a temporal relationship to the administration of the research intervention, follows a suspected pattern of response, or is otherwise logically related to the intervention, but an alternative cause is present.

## Unlikely

The adverse event is doubtfully related to the research intervention: the adverse event has a temporal or other relationship to the administration of the research intervention, but follows no known or suspected pattern of response, and an alternative cause is present.

#### Not Related

The adverse event is clearly NOT related to the research intervention: the adverse event has no temporal or other relationship to the administration of the research intervention, follows no known or suspected pattern of response, and an alternative cause is present.

#### 6.3 Serious Adverse Events

A serious adverse event (SAE) is any adverse event that:

- Results in death:
- Is life-threatening; the subject was at substantial risk of dying at the time of the adverse
  event, or use or continued use of the device or other medical product might have
  resulted in the death of the patient;
- Results in hospitalization (initial or prolonged);
- Results in disability or permanent damage; the event resulted in a substantial disruption of the person's ability to conduct normal life functions;
- Results in a congenital anomaly or birth defect;
- Requires intervention to prevent permanent impairment or damage; medical or surgical intervention was necessary to preclude permanent impairment of a body function, or prevent permanent damage to a body structure.
- Results in any other serious, important medical events; the event does not fit the other
  outcomes, but the event may jeopardize the patient and may require medical or surgical
  intervention to prevent one of the other outcomes.

In case of Serious Adverse Events (SAE), the Investigator must notify the Sponsor or its representative using the Adverse Event Form as soon as possible but at most within 24 hours of becoming aware of the event using the contact information below.

Sponsor Contact: Mukesh Ahuja E-mail: mahuja@medacta.us.com

Fax: (312) 546-6881

The Investigator should provide additional information on the SAE by updating the information on the Adverse Event Form and CRF as updates become available. The Sponsor may also ask for additional clinical reports including redacted source documents to be provided by the Investigator to assist in the assessment of the event. Significant new information and updates should continue to be submitted promptly to the Sponsor and entered on the Adverse Event CRF as they become available, and the Investigator should follow the SAE until it is resolved or no further improvement is expected.

New SAEs will only be documented for each patient until the last study-related clinic visit.

# 6.4 Unanticipated Adverse Device Effects

An UADE is defined as any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device/product, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the protocol or application, or any other unanticipated serious problem associated with a device/product that is related to the rights, safety, or welfare of subject. Adverse events that might reasonably occur because of placement or attempted placement of the product or during follow-up are identified through a risk assessment and summarized in the Instructions for Use.

If Medacta determines that a UADE presents an *unreasonable risk* to study subjects, Medacta will:

- terminate the investigation, or the parts of the investigation presenting that risk, within 5 working days after making the "unreasonable risk" determination, or within 15 working days of receiving notice of the UADE
- · immediately investigate and evaluate the adverse effect,
- report the results of the investigation to all reviewing IRBs and to all participating investigators within 10 working days after Medacta receiving notice of the UADE, and
- resume the study, if appropriate, as specified by the IRB.

# 6.5 Adverse Event Reporting

Adverse events should be reported to the overseeing IRB per the board's specified reporting requirements. The CRA or Sponsor's representative will review each IRB's reporting requirements with the site.

### 7 ETHICAL AND LEGAL ASPECTS

## 7.1 Institutional Review Board (IRB)

This trial can only be undertaken after full approval has been obtained through the IRB or Ethics Committee (EC). The approval(s) must cover the protocol and addenda, if applicable, as well as the Informed Consent Form, product brochure and manufacturer information (if applicable).

During the trial the following documents will be sent to the EC/IRB for their review:

- Changes to the product brochure and manufacturer information
- Reports of all Adverse Events that are rated serious, unexpected and associated with the study product and meet IRB reporting requirements.
- · All protocol amendments and revised Informed Consent Forms (if any).

For any protocol amendments that increase subject risk, the amendment and applicable Informed Consent Form revisions must promptly be submitted to the EC/IRB for review and approval prior to implementation of the change(s).

Reports on, and reviews of the trial and its progress will be submitted to the EC/IRB by the Investigator at intervals stipulated in their guidelines.

At the end of the trial, the Investigator will notify the EC/IRB about the trial completion.

## 7.2 Good Clinical Practice

This trial will be conducted in accordance with the current ICH-GCP-guidelines as specified for medical devices in ISO 14155.



Good Clinical Practice (GCP) is an international ethical and scientific quality standard for designing, conducting, recording and reporting trials that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety and well-being of trial subjects are protected, consistent with the principles that have their origin in the Declaration of Helsinki, and that the clinical trial data are credible.

#### 7.3 Informed Consent

Prior to entry in the study, the investigator must explain to potential subjects or their legal representatives the trial and the implications of participation. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not impact on the care the subject will receive for the treatment of his/her disease. Subjects will be told that alternative treatments are available if they refuse to take part and that such refusal will not prejudice future treatment. Finally, they will be told that competent authorities may access their records and authorized Sponsor's persons without violating the confidentiality of the subject, to the extent permitted by the applicable law(s) and/or regulations. By signing the Informed Consent Form (ICF) the subject or legally acceptable representative is authorizing such access.

The subject will be given sufficient time to read the informed consent form and to ask additional questions. After this explanation and before entry to the trial, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the Informed Consent must be given to the subject.

# 7.4 Confidentiality, Compliance, and Data Management

Provisions for maintaining and insuring (1) the confidentiality of data, subject records, and investigator information, (2) compliance with financial disclosure requirements, law, audit, debarment, (3) quality management system, (4) data management are set forth in the executed contract between Sponsor and participating clinical centers.

All HIPAA requirements for subject confidentiality will be maintained. All summary data shared beyond the Sponsor, Sponsor's representatives and the patients' clinical team will be deidentified. Such summary data will not contain any of the identifiable protected health information (PHI) listed below:

Data that includes any of the following identifiers are considered identifiable health information:

- Name
- Social Security number
- Medical Record Number
- Address by Street Location
- Address by Town/City/Zip Code
- Date of Birth
- Admission or Discharge Date
- Date of Death
- Telephone Number
- Fax Number
- Electronic E-Mail Address
- Web URLs
- Internet Protocol (IP) Address
- Health Plan Beneficiary Number
- Account Number
- Certificate/License Number
- Vehicle Identification Number and Serial Number, including License Plate Number

- Medical Device Identifiers and Serial Numbers
- Biometric Identifiers (finger and voice prints)
- Full Face Photographic Image
- · Any Other Identifier likely to identify the subject

### 8 SUBJECT DISCONTINUATION / WITHDRAWAL

Consent to participate in this study is completely voluntary. Consent may be withdrawn at any time, if desired by the study participant or the investigator may choose to discontinue the subject. Reasons for discontinuation of a patient from the clinical study may be (1) insufficient cooperation of the patient (non-compliance); (2) technical or administrative reasons (e.g., change of investigator or move of patient or cancelled/postponed surgery outside of window); or (3) death. To formally withdraw consent to participate in this study, the participant will need to notify their treating physician.

## 9 USE OF INFORMATION AND PUBLICATION

The information generated during this study is proprietary information and is considered the property of Medacta. This information cannot be used in publication without the written consent of Medacta.

# 10 References

- 1. Losina E, et al. Cost-effectiveness of Total Knee Arthroplasty in the United States: Patient Risk and Hospital Volume. *Arch Intern Med* (2009); 169(2):1113-1122.
- 2. Mont MA, et al. Single-Use Instruments, Cutting Blocks, and Trials Increase Efficiency in the Operating Room During Total Knee Arthroplasty: A Prospective Comparison of Navigated and Non-Navigated Cases. *J Arthroplasty* (2013); 28(7):1135-1140.
- Siegel Gw, et al. Cost Analysis and Surgical Site Infection Rates in Total Knee Arthroplasty Comparing Traditional vs. Single-Use Instrumentation. J Arthroplasty (2015); 30: 2271-2274
- 4. Lachiewicz PF, Henderson RA: Patient-specific Instruments for Total Knee Arthroplasty. J Am Acad Orthop Surg, (2013); 21:513-518.
- 5. Hetaimish BM, Khan MM, Simunovic N, Al-Harbi HH, Bhandari M, Zalzal PK. Meta-Analysis of Navigation vs Conventional Total Knee Arthroplasty. *J Arthroplasty* 27(6) 2012
- Kim YH, Kim JS, Choi Y, Kwon OR. Computer-Assisted Surgical Navigatoin Does Not Improve the Alignment and Orientation of the Components in Total Knee Arthroplasty. JBJS AM 91(1): 14-19, 2009
- Decking R, Markmann Y, Fuchs J, Puhl W, Scharf HP. Leg Axis After Computer-Navigated Total Knee Arthroplasty, A Prospective Randomized Trial Comparing Computer-Navigated and Manual Implantation. J Arthroplasty 20(3) 2005

- De Steiger RN, Liu YL, Graves SE. Computer navigation for total knee arthroplasty reduces revision rate for patients less than sixty-five years of age. JBJS Am 2015 Apr 15;97(8):635-42
- Johnson DR, Dennis DA, Kindsfater KA, Kim RH. Evaluation of Total Knee Arthroplasty Performed With and Without Computer Navigation: A Bilateral Total Knee Arthroplasty Study. J Arthroplasty 2013 28: 455-458
- Brown MJ, Matthews JR, Bayers-Thering MT, Phillips MJ, Krackow KA. Low Incidence of Postoperative Complications with Navigated Total Knee Arthroplasty. J Arthroplasty (2017) 1-7
- 11. Carter RE, Rush PF, Smid JA, Smith WL. Experience with Computer-Assisted Navigation for Total Knee Arthroplasty in a Community Setting. *J Arthroplasty* 23(5), 2008
- 12. Clayton AW, Cherian JJ, Banerjee S, Kapadia BH, Jauregui JJ, Harwin SF, Mont MA. Does the Use of Navigation in Total Knee Arthroplasty Affect Outcomes? *J Knee Surg* 2014; 27(3): 171-176
- Gholson JJ, Duchman KR, Otero JE, Pugely AJ, Gao Y, Callaghan JJ. Computer Navigated Total Knee Arthroplasty: Rates of Adoption and Early Complications. J Arthroplasty (2017) 1-7
- 14. Mont MA, Banerjee S. Navigation in Total Knee Arthroplasty: Truth, Myths, and Controversies. *Am J Orthop.* 2013 November; 42(11): 493-495